CLINICAL TRIAL: NCT05018364
Title: Serum Erythropoietin Level for Detection of Kidney and Brain Injuries in Asphyxiated Neonates in Neonatal Intensive Care Unit.
Brief Title: Serum Erythropoietin Level in Perinatal Asphyxia
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Ahmed Sayed, Doctor, Cairo University
Other Study IDs: MS-222-2020
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Perinatal Hypoxia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: measure serum erythropoietin level
  Interventions: Diagnostic Test: Serum erythropoietin level
- controls: measure serum erythropoietin level
  Interventions: Diagnostic Test: Serum erythropoietin level

INTERVENTIONS:
Diagnostic Test: Serum erythropoietin level — Evaluate serum erythropoietin level in neonates exposed to hypoxia compared to control group

SUMMARY:
This study is to evaluate brain and kidney injuries in full-term neonates with perinatal asphyxia by detecting specific biomarker in blood (Erythropoietin).

DETAILED DESCRIPTION:
Perinatal hypoxic-ischemic encephalopathy (HIE) is an important cause of brain injury in the newborn and can result in long-term devastating consequences. Acute kidney injury (AKI) occurs in (50 - 72%) among asphyxiated term infants. The kidney cells that make erythropoietin are sensitive to low oxygen levels in the blood that travels through the kidney. These cells make and release erythropoietin when the oxygen level is too low.

ELIGIBILITY:
Inclusion Criteria:

Cases group:

1. The presence of a sentinel hypoxic event immediately before or during delivery
2. History of fetal distress (bradycardia, late decelerations, absence of heart rate variability).
3. Need for neonatal resuscitation at delivery
4. One-min Apgar score <3 or 5-minApgar score<7
5. Metabolic acidosis (BE > 10 in cord blood)
6. Cardiocirculatory instability (CCI), clinical indications of hypoxic-ischemic encephalopathy (HIE) and multiple organ involvement (MOI).

Control group:

Newborns who were delivered normally after uncomplicated pregnancy. None of them have clinical nor biochemical signs of asphyxia.

Exclusion Criteria:

* Newborns who do not fulfill the above criteria.
* Newborns with congenital heart diseases and perinatal hemolytic anemia or congenital liver affection.
* Whose parents refuse to participate in the study.
* Cases above 4 days old.
* Preterm neonates (less than 37 weeks).

Ages: 1 Day to 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Data will be collected from full-term neonates (first 28 days of life) with perinatal hypoxia admitted in Neonatal Intensive Care Unit. Both sexes are included (males & females) .
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
correlation between serum erythropoietin level and brain injury | first 4 days of life
  measure level of serum erythropoietin by ELISA technique and test if can differentiate degree of brain hypoxia

CONTACTS AND LOCATIONS:
Overall Officials: Yosra Aboelnaga, Study Chair — Dryosra86@hotmail.com; Nermine Riad, Study Chair — docnermoo@gmail.com
Locations (1):
- faculty of medicine, Cairo university, Cairo, Egypt

REFERENCES:
- [Background] Sweetman DU, Onwuneme C, Watson WR, Murphy JF, Molloy EJ. Perinatal Asphyxia and Erythropoietin and VEGF: Serial Serum and Cerebrospinal Fluid Responses. Neonatology. 2017;111(3):253-259. doi: 10.1159/000448702. Epub 2016 Dec 1. PMID 27902983